CLINICAL TRIAL: NCT05690984
Title: Combination Post-transplant Consolidation Therapy With Isatuximab, Lenalidomide, Dexamethasone (IsaRD) in Multiple Myeloma Patients With Persistent Marrow Minimal Residual Disease (Elimination of MRD After Transplant; E-MAT)
Brief Title: Elimination of Minimal Residual Disease After Transplant
Acronym: EMAT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Anita D'Souza, Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00046592
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
Keywords: minimal residual disease; multiple myeloma; next-generation sequencing
MeSH Terms: conditions — Multiple Myeloma; Neoplasm, Residual | interventions — Dexamethasone; Calcium Dobesilate; isatuximab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Isatuximab in combination with lenalidomide and dexamethasone. (Experimental): The isatuximab, lenalidomide, and dexamethasone (IsaRD) therapy will be administered on an outpatient basis.
  Interventions: Drug: Dexamethasone; Drug: Isatuximab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone will be used for the double purpose of premedication and therapeutic effect. On Day 1 of Cycle 1, subjects will be administered 40 mg dexamethasone as an IV infusion. On Days 8, 15, 22 of Cycle 1 and Days 1 and 15 of Cycles 2-4, dexamethasone will be given as a single oral dose of 40 mg. For Cycles 5-12, dexamethasone will be given as a single oral dose of 4 mg on Days 1 and 15.
  Other Names: Decadron; Dexasone; Diodex; Hexadrol; Maxidex
Drug: Isatuximab — Following premedication (if applicable), subjects will be given isatuximab 10 mg/kg body weight as an intravenous (IV) infusion on Days 1, 8, 15, and 22 (i.e., weekly) during Cycle 1 and on Days 1 and 15 (i.e., Q2W) during Cycles 2-12.
  Other Names: Sarclisa
Drug: Lenalidomide — On Days 1-21 for all 12 cycles, lenalidomide will be given to subjects as a single daily oral dose.
  Other Names: Revlimid

SUMMARY:
This is a single-center, single-arm, phase II study that will enroll multiple myeloma (MM) patients with persistent bone marrow minimal residual disease (MRD) post autologous stem cell transplant (ASCT) irrespective of the International Myeloma Working Group (IMWG) response.

DETAILED DESCRIPTION:
Thirty-one study subjects will be enrolled at Froedtert Hospital and the Medical College of Wisconsin Cancer Center. Enrolled subjects will receive a combination of isatuximab, lenalidomide, and dexamethasone (IsaRD) for 12 28-day cycles. The primary objective of this study is to determine bone marrow (BM) MRD ≤1x10^5 negativity rate, as measured by the clonoSEQ® next-generation sequencing (NGS) assay, at the end of 12 months of IsaRD treatment. Other objectives will further assess efficacy, tolerability, and molecular response to the IsaRD regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Eastern Cooperative Oncology Group (ECOG) Performance Status criteria of 0-2.
3. Must have archival bone marrow sample at time of diagnosis that can be used for clonality identification for NGS if not already performed.
4. Presence of residual bone marrow minimal residual disease (MRD) positivity by clonoSEQ® next-generation sequencing (NGS) 90-120 days post autologous stem cell transplantation.
5. Histologically confirmed diagnosis of symptomatic multiple myeloma (patients with multiple myeloma with secondary amyloidosis are eligible, but no amyloid treatment will be allowed while on study).
6. Received autologous stem cell transplant as upfront therapy for myeloma (defined as ASCT within one year of diagnosis of symptomatic MM).
7. Adequate organ function as defined below:

   * Absolute neutrophil count (ANC) ≥1,000/mm^3.
   * Platelet count ≥75,000/mm^3; platelet transfusions to help patients meet eligibility criteria are not allowed within seven days before study enrollment.
   * Total bilirubin ≤1.5 x the upper limit of the normal range (ULN)
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 x ULN
8. Pregnancy It is not known what effects this treatment has on human pregnancy or development of the embryo or fetus. Therefore, female subjects participating in this study should avoid becoming pregnant, and male subjects should avoid impregnating a female partner. Non-sterilized female subjects of reproductive age and male subjects should use effective methods of contraception through defined periods during and after study treatment as specified below.

   Female participants: A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:
   * Not a female of childbearing potential (FCBP), OR
   * A FCBP who must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10-14 days prior to and again within 24 hours prior to starting study medication and before each cycle of study treatment and must either commit to continue abstinence from heterosexual intercourse or apply a highly effective method of birth control during the intervention period and for at least five months after the last dose of isatuximab treatment Male participants: A male participant, even if surgically sterilized (i.e., status post-vasectomy), must agree to use contraception during the intervention period and for at least five months after the last dose of isatuximab treatment and refrain from donating sperm during this period.
9. All study participants must be registered into the mandatory Revlimid REMS® program and be willing to comply with its requirements.
10. Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

1. Evidence of MM disease progression any time prior to enrollment.
2. Administration or planned administration of any other concomitant chemotherapy, immunotherapy, or any ancillary therapy that would be considered a treatment of multiple myeloma from Day +30 post-transplant through discontinuation from study. Local radiation therapy is allowed. Subjects may be on corticosteroids if they are being given for disorders other than multiple myeloma (e.g., adrenal insufficiency, rheumatoid arthritis, etc.)
3. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
4. Prior organ transplant requiring immunosuppressive therapy.
5. Known to be human immunodeficiency virus (HIV) positive.
6. Known to have hepatitis A, B, or C active infection. If hepatitis positive, patient may still be per the notes below.

   • Uncontrolled or active hepatitis B virus (HBV) infection: Patient with positive HBsAg and/or HBV DNA.

   Of Note:
   * Patient can be eligible if anti-HBc IgG positive (with or without positive anti-HBs) but HBsAg and HBV DNA are negative.
   * If anti-HBV therapy in relation with prior infection was started before initiation of investigational medicinal product, the anti-HBV therapy and monitoring should continue throughout the study treatment period.
   * Patient with negative HBsAg and positive HBV DNA observed during screening period will be evaluated by a specialist for start of anti-viral treatment: study treatment could be proposed if HBV DNA becomes negative and all the other study criteria are still met.

     * Active hepatitis C virus (HCV) infection: positive HCV RNA and negative anti-HCV.

   Of Note:
   * Patients with antiviral therapy for HCV started before initiation of investigational medicinal product and positive HCV antibodies are eligible. The antiviral therapy for HCV should continue throughout the treatment period until seroconversion.
   * Patients with positive anti-HCV and undetectable HCV RNA without antiviral therapy for HCV are eligible.
7. Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
8. Concurrent hematologic or non-hematologic malignancy requiring treatment (other than multiple myeloma and secondary amyloidosis).
9. Cardiac syncope, uncompensated New York Heart Association (NYHA) Class 3 or 4 congestive heart failure, myocardial infarction within the previous six months, unstable angina pectoris, clinically significant repetitive ventricular arrhythmias despite antiarrhythmic treatment, severe orthostatic hypotension, or clinically important autonomic disease.
10. Major surgery within 14 days prior to start of study treatment (Note: vertebroplasty and kyphoplasty are not considered major surgery).
11. Infection requiring systemic antibiotic therapy or other serious infection within 14 days prior to start of study treatment.
12. Participation in other clinical trials, including those where a subject received an investigational drug within 30 days or five half-lives of the investigational drug prior to start of study treatment, whichever is longer.
13. Any clinically significant, uncontrolled medical conditions that, in the investigator's opinion, would expose the subject to excessive risk or may interfere with compliance or interpretation of the study results.
14. Hypersensitivity or history of intolerance to steroids, mannitol, pregelatinized starch, sodium stearyl fumarate, histidine (as base and hydrochloride salt), arginine hydrochloride, poloxamer 188, sucrose or any of the other components of study intervention that are not amenable to premedication with steroids and H2 blockers or would prohibit further treatment with these agents.
15. Pregnant or breastfeeding subjects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
The number of subjects who have less than MRD. | One year
  Bone marrow MRD negative at a cutoff sensitivity of ≤1x10^5 sequence copies as measured by the clonoSEQ® next-generation sequencing assay at the end of IsaRd treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Meera Mohan, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No